CLINICAL TRIAL: NCT01697293
Title: A Phase I-II Study of PTX-200 Plus Sequential Weekly Paclitaxel Followed by Dose-Dense Doxorubicin and Cyclophosphamide in Patients With Metastatic and Locally Advanced Breast Cancer
Brief Title: PTX-200, Paclitaxel, Doxorubicin Hydrochloride, and Cyclophosphamide in Treating Patients With Stage IIB-IV Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: criteria for continuing enrollment in Phase 2 portion was not met
Sponsor: Prescient Therapeutics, Ltd. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-269; NCI-2013-01311 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-051; TCN-PM; PTX-200-BC-1501.1; PTX-200; 007884; 2011-269 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH); R01CA098473 (NIH)
Record Dates: First submitted 2012-09-13; First posted 2012-10-02 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Breast Adenocarcinoma; Estrogen Receptor Positive; HER2/Neu Negative; Recurrent Breast Carcinoma; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Paclitaxel; Taxes; triciribine phosphate; triciribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, surgery) (Experimental): COURSES A 1-12 (PHASE I & II): Patients receive triciribine phosphate IV over 60 minutes on days 1, 8, and 15, 29, 36, 43, 57, 64, and 71 and paclitaxel IV over 1 hour on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 79. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  COURSES B 1-4 (PHASE II): Patients receive doxorubicin hydrochloride IV over 5-10 minutes and cyclophosphamide IV over 30-60 minutes on day 1. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  SURGERY (PHASE II): Eligible patients undergo modified radical mastectomy, radical mastectomy, segmental mastectomy or lumpectomy with an axillary lymph node dissection or biopsy.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Procedure: Therapeutic Conventional Surgery; Drug: Triciribine Phosphate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Therapeutic Conventional Surgery — Undergo modified radical mastectomy, radical mastectomy, segmental mastectomy or lumpectomy with an axillary lymph node dissection or biopsy
Drug: Triciribine Phosphate — Given IV
  Other Names: 1, 5-Dihydro-5-methyl-1-(5-O-phosphono-.beta.-D-ribofuranosyl)-1,4,5, 6,8-pentaazaacenaphthylen-3-amine; 1,4, 5,6,8-Pentaazaacenaphthylen-3-amine, 1, 5-dihydro-5-methyl-1-(5-O-phosphono-.beta.-D-ribofuranosyl)- (9CI); 1,4,5,6, 8-Pentaazaacenaphthalen-3-amine, 1, 5-dihydro-5-methyl-1-(5-O-phosphono-.beta.-D-ribofuranosyl)-; 3-Amino-1, 5-dihydro-5-methyl-1-.beta.-D-ribofuranosyl-1,4,5,6, 8-pentaazaacenaphthylene 5'-(dihydrogen phosphate); TCN; Triciribine; Tricycloside Phosphate

SUMMARY:
This phase I/II trial studies the side effects and the best dose of triciribine phosphate when given together with paclitaxel, doxorubicin hydrochloride, and cyclophosphamide and to see how well they work in treating patients with stage IIB-IV breast cancer. Triciribine phosphate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel, doxorubicin hydrochloride, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving triciribine phosphate with paclitaxel, doxorubicin hydrochloride, and cyclophosphamide may be a better treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose of PTX-200 (triciribine phosphate) given on days 1, 8, and 15 every 28 days (maximum of 9 doses) when combined with weekly paclitaxel (80 mg/m^2) for 12 weeks in patients with metastatic breast cancer. (Phase I and Expansion Cohort) II. To determine the pathologic response rate (Residual Cancer Burden [RCB] score 0-1) after sequential weekly paclitaxel plus PTX 200 weekly, 3 weeks out of 4, followed by doxorubicin (doxorubicin hydrochloride) (60 mg/m^2) and cyclophosphamide (600 mg/m^2) every 2 weeks x 4 cycles in patients with clinical stage IIB-IIIC breast cancer. (Phase II).

III. To determine the feasibility and safety of the combination of sequential weekly paclitaxel plus PTX-200 (days 1, 8, and 15) followed by doxorubicin/cyclophosphamide. (Phase II)

SECONDARY OBJECTIVES:

I. To correlate pre-treatment levels of erb-b2 receptor tyrosine kinase (ErbB)1, 2, 3, 4 and zinc finger protein 217 (ZNF217), and phosphorylated levels of v-akt murine thymoma viral oncogene homolog 1 (Akt), signal transducer and activator of transcription 3 (acute-phase response factor) (STAT3), extracellular signal-regulated protein kinases 1 and 2 (Erk1/2) to pathologic (RCB score 0-1) response (Sebti laboratory [lab]). (Phase I or II) II. To correlate the percent decrease in the levels of phosphorylated (phospho-)Akt (S473), phospho-S6 (S235-236), phospho-proline-rich Akt substrate, 40 kDa (PRAS40) (threonine [Thr]246), phosphatase and tensin homolog (PTEN), Stathmin, pyruvate dehydrogenase kinase, isozyme 1 (PDK1), cyclin D1, phospho-STAT3, ras homolog gene family, member C (Rho C), and phospho-Erk 1-2 with pathologic response rate (RCB score 0-1), percent inhibition of proliferation (Ki-67) and percent induction of apoptosis (terminal deoxynucleotidyl transferase dUTP nick end labeling [Tunel]) (Sebti lab). (Phase I or II)

OUTLINE: This is a phase I, dose-escalation study of triciribine phosphate followed by an expansion cohort and a phase II study.

COURSES A 1-12 (PHASE I & II): Patients receive triciribine phosphate intravenously (IV) over 60 minutes on days 1, 8, and 15, 29, 36, 43, 57, 64, and 71 and paclitaxel IV over 1 hour on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 79. Treatment repeats every week for 12 courses in the absence of disease progression or unacceptable toxicity.

COURSES B 1-4 (PHASE II): Patients receive doxorubicin hydrochloride IV over 5-10 minutes and cyclophosphamide IV over 30-60 minutes on day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.

SURGERY (PHASE II): Eligible patients undergo modified radical mastectomy, radical mastectomy, segmental mastectomy or lumpectomy with an axillary lymph node dissection or biopsy.

After completion of study treatment, patients with metastatic disease are followed up every 3 months for 1 year and patients with locally advanced disease are followed up every 6 months for 2 years and then yearly for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Phase I and expansion cohort: Patients must have histologically or cytologically confirmed adenocarcinoma of the breast associated with clinical stage: IV (see American Joint Committee on Cancer [AJCC] staging criteria, 7th edition) or stage IIB-IIIC (expansion cohort only)
* Phase II: Patients must have histologically or cytologically confirmed adenocarcinoma of the breast associated with the following clinical stage: IIB, IIIA, IIIB, or IIIC (see AJCC staging criteria, 7th edition); the tumor must be human epidermal growth factor receptor 2 (Her2)/neu negative (by DAKO HercepTest, fluorescence based in situ hybridization [FISH], or other approved assay)
* Phase I and expansion cohort: Up to two prior non-taxane chemotherapy regimens for metastatic disease are permitted for patients enrolled on the phase I portion of the trial; patients with HER2/neu positive breast cancer are not eligible; patients treated with prior anthracycline therapy as neoadjuvant, adjuvant, or metastatic therapy are not eligible unless the following conditions are met: (a) prior cumulative doxorubicin dose is =< 240 mg/m^2 (or epirubicin dose is =< 400 mg/m^2), and (b) left ventricular ejection fraction (LVEF) obtained at baseline is at least 50% (or >= 5% above lower institutional limits of normal whichever is higher); patients with estrogen receptor (ER)-positive disease are required to have relapse or progression on at least one line of endocrine therapy
* Phase II: No prior chemotherapy, irradiation, or definitive therapeutic surgery (e.g., mastectomy or lumpectomy or axillary dissection) for this malignancy; patients who have had a prior sentinel lymph node biopsy for this malignancy are eligible
* Patients who received tamoxifen or another selective estrogen receptor modulator (SERM) for prevention or treatment of breast cancer or for other indications (e.g., osteoporosis, prior ductal carcinoma in situ [DCIS]), or who receive aromatase inhibitors for prevention or treatment of breast cancer, are eligible; patients who are hormone-receptor positive and who have received other hormonal agents for the treatment of breast cancer (e.g., Fulvestrant) are also eligible; tamoxifen therapy or other hormonal agents should be discontinued at least 1 week before the patient is enrolled on this study
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Leukocytes >= 3,000/uL
* Absolute neutrophil count =< 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal
* Left ventricular ejection fraction (LVEF) within normal institutional limits
* Creatinine within normal institutional limits
* LVEF at or above institutional lower limits of normal (>= 50%), or at least 5% above lower limits of normal if prior anthracycline exposure (by echocardiogram or nuclear scan within 12 weeks of registration)
* Electrocardiogram (ECG) corrected QT (QTC) < 450 msec
* Serum calcium within normal institutional limits
* Serum phosphorus within normal institutional limits
* Fasting glucose within normal limits
* Patients must be disease-free of prior invasive malignancies for >= 2 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix (for phase II only); patients with the following prior or concurrent diagnoses are eligible: lobular carcinoma in situ, contralateral ductal carcinoma in situ, or contralateral invasive ductal and/or lobular cancer (and no prior adjuvant chemotherapy for previous breast malignancy)
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents during protocol therapy, or up to 30 days prior to beginning protocol therapy; there should be a least a 1-week interval between last dose of endocrine therapy and protocol therapy, and at least 3 weeks for the last dose of biologic therapy (eg, bevacizumab) or cytotoxic therapy (or 2 weeks for capecitabine or weekly paclitaxel, 6 weeks for mitomycin-C and nitrosoureas), and adequately recovered from adverse effects from prior therapy to meet all other eligibility criteria
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PTX-200 or other agents used in the study (e.g., imidazoles, quinolones)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, diabetes mellitus requiring therapy (insulin or oral hypoglycemic agents), congenital prolonged QT syndrome, requirement for a drug known to prolong the QT interval, a history of QT prolongation, a screening QTc >= 450 msec, hypertriglyceridemia requiring therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with PTX-200; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients receiving combination antiretroviral therapy are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Pathologic response (RCB score 0-1), assessed using the criteria of Chevallier (Phase II) | At time of surgery
  The estimated pCR along with exact confidence interval will be presented.
Recommended phase II dose of triciribine phosphate, based on the incidence of dose-limiting toxicity graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (Phase I) | 28 days
  Adverse effects will be summarized using frequency tables. The proportion of patients who completed all 12 courses of paclitaxel (at full dose or with dose modification) will be tabulated.

SECONDARY OUTCOMES:
Clinical complete response and partial response, based on tumor measurements obtained by physical exam | Up to 20 weeks (completion of courses B 1-4)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sparano, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - Albert Einstein College of Medicine, The Bronx, New York